CLINICAL TRIAL: NCT07129343
Title: A Clinical Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Recombinant Von Willebrand Factor (rVWF) With or Without ADVATE in the Treatment of Bleeding Episodes in Chinese Subjects Diagnosed With Von Willebrand Disease
Brief Title: A Study of Recombinant Von Willebrand Factor (rVWF) in Chinese Participants With Von Willebrand Disease (vWD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-577-3002
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Von Willebrand Disease (VWD)
Keywords: Drug Therapy
MeSH Terms: conditions — von Willebrand Diseases | interventions — Factor VIII; F8 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All Participants With VWD (Experimental): Participants will receive a single intravenous (IV) dose of VONVENDI at baseline PK assessment. During the 12-month on-demand (OD) treatment period, any bleeding episodes requiring replacement therapy with VWF will be treated with VONVENDI with or without ADVATE. Participants may also receive VONVENDI with or without ADVATE intravenous infusions, when indicated deemed necessary for perioperative bleeding management [major, minor and oral surgery]. Participants will receive initial dose of VONVENDI of 40 to 80 IU/kg of body weight.
  Interventions: Biological: VONVENDI; Biological: ADVATE

INTERVENTIONS:
Biological: VONVENDI — VONVENDI is administered by intravenous injection.
  Other Names: vonicog alfa; TAK-577; rVWF
Biological: ADVATE — ADVATE is administered by intravenous injection.
  Other Names: rFVIII; Octocog alfa

SUMMARY:
The main aim of this study is to find out if VONVENDI is safe for adult Chinese participants with VWD. The study will also check how well VONVENDI helps control bleeding with or without product ADVATE in the participants who may need elective surgery or dental procedures. In addition, the study will also examine how VONVENDI is processed by the body (known as pharmacokinetic [PK]) and how the drug helps the body respond or improve a condition (pharmacodynamic [PD]).

Participants will receive an initial dose of VONVENDI of 40 to 80 international units per kilogram (IU/kg) of body weight. If a participant's baseline factor VIII (FVIII) level is not high enough to help stop bleeding, VONVENDI will be given along with 30 to 45 IU/kg of ADVATE rFVIII.

Participants will be in the study for approximately 14 months. During the study, participants will be followed up at clinics or over telephone calls.

ELIGIBILITY:
Inclusion Criteria

1. Participant must voluntarily sign an institutional review board (IRB)/independent ethics committee-approved written informed consent form after all relevant aspects of the study have been explained and discussed with the participant.
2. Participant has a documented diagnosis of severe VWD (baseline VWF:RCo less than [<]20 international units [IU]deciliter [dL]) with a diagnosis of VWD type verified per the following recommended criteria:

   * Type 1 (von Willebrand factor:Ristocetin cofactor activity [VWF:RCo] <20 IU/dL and by VWF activity/VWF:antigen [Ag] ratio) or,
   * Type 2A or type 2B (by VWF activity/VWF:Ag ratio and multimer pattern, with genetics if necessary), type 2N (FVIII:C <10% and genetics), type 2M (by VWF activity/VWF:Ag ratio and multimer pattern) or
   * Type 3 (VWF:Ag <=3 IU/dL). Diagnosis is confirmed, when applicable, by genetic testing and/or by multimer analysis.
3. Participant is at least 18 years of age at screening.
4. Participant is ethnic Chinese and lives in China, including those from Taiwan, Hong Kong, and Macao.
5. If female of childbearing potential, participant presents with a negative pregnancy test and agrees to employ adequate birth control measures for the duration of the study.
6. Participant is willing and able to comply with the requirements of the protocol.
7. Participant has had a minimum of 3 documented bleeds that indicated the need for VWF coagulation factor replacement therapies during the previous 12 months prior to enrollment.

Exclusion Criteria

1. Participant has been diagnosed with pseudo VWD or another hereditary or acquired coagulation disorder other than VWD (example [eg], qualitative and quantitative platelet disorders or elevated prothrombin time [PT]/international normalized ratio >1.4).
2. Participant has a history or presence of a VWF inhibitor at screening.
3. Participant has a documented history of a VWF:RCo half-life of <6 hours.
4. Participant has a history or presence of a FVIII inhibitor with a titer greater than or equal to [>=] 0.6 Bethesda units per milliliter [BU/mL] (by Bethesda assay or Bethesda method with Nijmegen modification).
5. Participant has a known hypersensitivity to any of the components of the study drugs, such as to mouse or hamster proteins.
6. Participant has a medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis, mild asthma, food allergies or animal allergies.
7. Participant has a medical history of a thromboembolic event.
8. Participant is human immunodeficiency virus (HIV) positive with an absolute cluster of differentiation 4 (CD4) count <200/cubic millimeter (mm^3).
9. Participant has been treated with an immunomodulatory drug, other than antiretroviral chemotherapy eg, α-interferon, or corticosteroid agents at a dose equivalent to hydrocortisone greater than 10 milligram (mg)/day (excluding topical treatment [eg, ointments, nasal sprays]), within 30 days prior to signing the informed consent (or assent, if appropriate).
10. Participant is pregnant or lactating at the time informed consent is obtained.
11. Participant has participated in another clinical study involving an IP, or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
12. Participant is diagnosed with progressive fatal disease and/or has a life expectancy of less than 15 months.
13. Participant is member of the study team conducting this study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (that is, children, partner/spouse, siblings, parents) as well as employees.
14. Participant has an acute illness (eg, influenza, flu-like syndrome, allergic rhinitis/conjunctivitis, nonseasonal asthma) at screening.
15. Participant is diagnosed with significant liver disease, as evidenced by, but not limited to, any of the following: serum alanine aminotransferase (ALT) greater than 5 times the upper limit of normal; hypoalbuminemia; portal vein hypertension (eg, presence of otherwise unexplained splenomegaly, history of esophageal varices) or liver cirrhosis classified as Child-Pugh class B or C.
16. Participant has been diagnosed with renal disease, with a serum creatinine level >=2.5 milligram per deciliter (mg/dL).
17. Participant has a platelet count <100,000/ milliliter (mL) at screening (except for participants with type 2B VWD, whose platelet count[s] at screening will be evaluated taking into consideration historical trends in platelet counts and the investigator's medical assessment of the participant's condition).
18. Participant has cervical or uterine conditions causing menorrhagia or metrorrhagia (including infection, dysplasia).
19. In the judgment of the investigator, the participant has another clinically significant concomitant condition (eg, uncontrolled hypertension) that may pose additional risks for the participant.
20. Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-11-25 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 14 months
  A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. An SAE is any untoward medical occurrence that at any dose: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event in the opinion of the healthcare provider, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above. TEAEs consist of both serious and non-serious adverse events.
Number of Participants With TEAEs by Severity | Up to 14 months
  Number of participants with severity of TEAE will be reported.
Number of Participants With TEAEs and SAEs by Causality | Up to 14 months
  Number of participants with causality related TEAEs and SAEs will be reported.
Number of Participants With Thromboembolic Events and Severe Hypersensitivity Reactions | Up to 14 months
  Number of participants with thromboembolic events and severe hypersensitivity reactions will be reported.
Number of Participants Who Develop Neutralizing (Inhibitory) Antibodies to VWF and FVIII | Up to 14 months
  Number of participants who develop neutralizing antibodies to VWF and FVIII will be reported.
Number of Participants Who Develop Binding Antibodies to VWF and FVIII | Up to 14 months
  Number of participants who develop total binding antibodies to VWF and FVIII will be reported.
Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters | Up to 14 months
  Number of participants with clinically significant abnormalities from baseline values in laboratory parameters per investigator assessment will be reported.
Number of Participants With Clinically Significant Abnormalities in 12-lead Electrocardiogram (ECG) | Up to 14 months
  Number of participants with clinically significant abnormalities from baseline values in ECG per investigator assessment will be reported.
Number of Participants With Clinically Significant Abnormalities in Vital Signs Parameters | Up to 14 months
  Number of participants with clinically significant abnormalities from baseline values in vital sign parameters per investigator assessment will be reported.

SECONDARY OUTCOMES:
Number of Infusions of VONVENDI With or Without ADVATE per Bleeding Episode | Up to 12 months
  Number of infusions of VONVENDI with or without ADVATE per bleeding episode will be reported.
Number of Infusions of ADVATE per Bleeding Episode | Up to 12 months
  Number of infusions of ADVATE per bleeding episode will be reported.
Weight-adjusted Consumption of VONVENDI and ADVATE per Bleeding Episode | Up to 12 months
  Weight-adjusted consumption of VONVENDI and ADVATE per bleeding episode will be reported.
Time to Resolution of Bleeding Episodes | Up to 12 months
  Time to resolution of the bleeding episodes will be calculated as the difference between the date/time of the first IP infusion for the bleeding episode to the date/time of the bleeding episode resolution.
Area Under the Plasma Concentration/Time Curve From Time 0 to Infinity (AUC0-inf) for VWF: Ristocetin Cofactor (VWF:Rco), VWF: Antigen (VWF:Ag) and VWF: Collagen Binding Capacity (VWF:CB) | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  AUC0-inf parameter at the baseline PK assessment will be calculated using noncompartmental analysis (NCA) for VWF:RCo, VWF:Ag, and VWF:CB.
Dose Normalized AUC (0-inf) for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Dose normalized AUC0-inf parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
AUC From Time 0 to 96 Hours (AUC0-96h) for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  AUC0-96h parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Dose Normalized AUC(0-96h) for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Dose normalized AUC0-96h parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Maximum Plasma Concentration (Cmax) for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Cmax parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Dose Normalized Cmax for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Dose normalized Cmax parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Time to Reach Maximum Plasma Concentration (Tmax) for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Tmax parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Mean Residence Time for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Mean residence time parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Clearance for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Clearance parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Terminal Half-life (T1/2) for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  T1/2 parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Volume of Distribution at Steady State (Vss) for VWF:RCo, VWF:Ag and VWF:CB | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Vss parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo, VWF:Ag, and VWF:CB.
Incremental Recovery (IR) at Cmax for VWF:RCo and VWF:Ag | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  IR parameter at the baseline PK assessment will be calculated using NCA for VWF:RCo and VWF:Ag.
AUC From Time 0 to Last time of Measurable Activity (AUC0-tlast) for Factor VIII:Coagulation Activity (FVIII:C) | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  AUC0-tlast parameter at the baseline PK assessment will be calculated using NCA for FVIII: C.
Dose Normalized AUC0-tlast for FVIII:C | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Dose Normalized AUC0-tlast parameter at the baseline PK assessment will be calculated using NCA for FVIII: C.
AUC0-96h for FVIII:C | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  AUC0-96h parameter at the baseline PK assessment will be calculated using NCA for FVIII: C.
Dose Normalized AUC0-96h for FVIII:C | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Dose normalized AUC0-96h parameter at the baseline PK assessment will be calculated using NCA for FVIII: C.
Cmax for FVIII:C | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Cmax parameter at the baseline PK assessment will be calculated using NCA for FVIII: C.
Dose Normalized Cmax for FVIII:C | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Dose Normalized Cmax parameter at the baseline PK assessment will be calculated using NCA for FVIII: C.
Tmax for FVIII:C | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Tmax parameter at the baseline PK assessment will be calculated using NCA for FVIII: C.
Plasma Level of VONVENDI based on Von Willebrand Factor: Ristocetin Cofactor (VWF:Rco) | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Plasma level of VONVENDI based on VWF:Rco will be reported.
Plasma Level of VONVENDI based on Von Willebrand Factor Antigen (VWF:Ag) | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Plasma level of VONVENDI based on VWF:Ag will be reported.
Plasma Level of VONVENDI based on Von Willebrand Factor Collagen Binding (VWF:CB) | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Plasma level of VONVENDI based on VWF:CB will be reported.
Plasma Level of Factor VIII Clotting (FVIII:C) | At baseline: Within 1 hour pre-infusion, 0.25, 0.50, 1, 3, 6, 12, 24, 30, 48, 72, and 96 hours post-infusion
  Plasma level of FVIII:C will be reported.
Total Hemostatic Efficacy Assessment 24 hours After Last Perioperative IP Infusion or at Day 14 Postoperative Visit | At 24 hours or Day 14
  The overall hemostatic efficacy of VONVENDI, with or without ADVATE, will be assessed by the investigator using the hemostatic efficacy assessment rating scale either 24 hours after the last perioperative infusion or at the Day 14 postoperative visit, whichever comes first.
Total Volume of Actual and Predicted Intraoperative Blood Loss After the Surgery as Assessed by the Operating Surgeon | From Intraoperative through completion of surgery (up to Day 14)
  Intraoperative actual blood loss will be assessed by the operating surgeon at the completion of surgery using a predefined 4-point rating scale. 1- Excellent (intraoperative blood loss was less than or equal to the maximum expected for the type of procedure performed in a hemostatically normal individual [<=]100 percent [%]); 2- Good (intraoperative blood loss up to 50% more than the maximum expected blood loss for the type of procedure performed in a hemostatically normal individual [101%-150%]); 3- Moderate (intraoperative blood loss exceeding 50% of the expected for the type of procedure performed in a hemostatically normal individual [greater than (>)150%]); 4- None (uncontrolled hemorrhage due to an inadequate therapeutic response despite appropriate dosing, necessitating a change of clotting factor replacement regimen). Lower scores indicate better hemostatic efficacy. Scoring is calculated by comparing the actual blood loss versus predicted blood loss.
Intraoperative Hemostatic Efficacy Score as Assessed by Operating Surgeon at Completion of Surgery | At completion of surgery (up to Day 14)
  The hemostasis assessment rating scale ranges from 1 to 4, where 1 = Excellent, 2 = Good, 3 = Moderate, and 4 = None. Lower scores indicate better hemostatic efficacy.
Daily Intra- and Postoperative Weight-adjusted Dose of VONVENDI With or Without ADVATE Through Postoperative Day 14 | From day of surgery through postoperative Day 14
  Daily intra- and postoperative weight-adjusted dose of VONVENDI with or without ADVATE through postoperative day 14 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing
  - Nanfang Hospital Southern Medical University, Guangzhou
  - Jinan Central Hospital, Jihan
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/bf56bcc8ebb94107??page=1&idFilter=TAK-577-3002